CLINICAL TRIAL: NCT06848595
Title: Effects of Dexmedetomidine Versus Magnesium Sulfate on Cerebral Oxygen Saturation During Spine Surgery: a Prospective Randomized Controlled Study
Brief Title: Mg Sulfate Versus Dexmedetomidine on Cerebral Oxygen Saturation
Acronym: mg/dex/rSO2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ibrahim Elsayed, doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36265MD317/11/24
Record Dates: First submitted 2025-02-21; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Desaturation Events; Spine Surgeries
MeSH Terms: interventions — Magnesium Sulfate; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MgSO4 (Active Comparator): loading dose of 40 mg/kg of magnesium sulfate diluted in 50 ml of 0.9% saline IVI will be given in 10 min before anesthesia induction then continuous infusion of 10 mg/kg/hour during the surgery.
  Interventions: Procedure: spine surgery; Drug: Magnesium sulfate
- dex. (Active Comparator): Patients will receive loading dose of 1 mcg/kg dexmedetomidine diluted in 50 ml of saline 0.9% IVI will be given in 10 min before anesthesia induction then continuous infusion of 0.5 mcg/kg/hour during the surgery.
  Interventions: Procedure: spine surgery; Drug: Dexmedetomidine
- control (Placebo Comparator): Patients will receive the same volume of normal saline.
  Interventions: Procedure: spine surgery; Drug: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Procedure: spine surgery — spine surgery in prone position
Drug: Magnesium sulfate — Patients will receive loading dose of 40 mg/kg of magnesium sulfate diluted in 50 ml of 0.9% saline IVI will be given in 10 min before anesthesia induction then continuous infusion of 10 mg/kg/hour during the surgery.
  Arms: MgSO4
Drug: Dexmedetomidine — Patients will receive loading dose of 1 mcg/kg dexmedetomidine diluted in 50 ml of saline 0.9% IVI will be given in 10 min before anesthesia induction then continuous infusion of 0.5 mcg/kg/hour during the surgery.
  Arms: dex.
Drug: Normal Saline (0.9% NaCl) — Patients will receive the same volume of normal saline.
  Arms: control

SUMMARY:
This study is to evaluate the effects of dexmedetomidine and magnesium sulfate on cerebral oxygen saturation in patients undergoing spine surgeries as adjuvant to general anesthesia guided by cerebral oximetry. The main aims to are Incidence of cerebral desaturation events and duration of cerebral desaturation events.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 60 years old.
* either gender.
* American Society of Anesthesiologists (ASA) physical status I and II.

Exclusion Criteria:

* Patient refusal to participate in research.
* History of preoperative neuromuscular disease.
* Patients with preexisting cerebral pathology (such as previous episodes of cerebral ischemia or stroke).
* History of psychiatric illness.
* History of orthostatic hypotension, myocardial infarction, uncontrolled hypertension or documented carotid stenosis.
* Coagulopathy disorder.
* Patients receiving magnesium supplementation.
* Chronic use of opioids.
* Current treatment with a β-blocker or calcium channel blocker.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-23 (Estimated); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of cerebral desaturation events. | intraoperative

SECONDARY OUTCOMES:
Duration of cerebral desaturation events | intraoperative
change in heart rate in beats | intraoperative
change in blood pressure in mmHg | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Said Elgebaly, professor, Study Director — Tanta University; Shimaa Farouk Abdelkader, professor, Study Director — Tanta University

IPD SHARING:
Plan to Share IPD: No